CLINICAL TRIAL: NCT05550064
Title: Evaluating Effects of Prepartum Structured Contraceptive Counseling to Increase Postpartum Use of Long-acting Reversible Contraception
Brief Title: Structured Contraceptive Counseling During Pregnancy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dalarna University (Other)
Responsible Party: Principal Investigator, Niklas Envall, PhD, RNM, Senior Lecturer, Dalarna University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SPR1
Record Dates: First submitted 2022-09-15; First posted 2022-09-22 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Contraception; Intrauterine Device; Contraceptive Implant; Long-acting Reversible Contraception; Counseling

STUDY DESIGN:
Intervention Model Description: Pregnant women will receive an intervention for structured contraceptive counseling from participating clinics. Follow-up will be through e-surveys at 6, 12, 18, and 24 months postpartum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention arm (Experimental): Evidence-based intervention for SCC, previously evaluated in a cluster randomized trial (doi:10.1111/1471-0528.16754) The intervention for prepartum SCC will consist of four different parts, adjusted to suit pregnant women with emphasis on immediate start when applicable:
  1. An educational video presenting available contraceptive methods
  2. 4 Key questions concerning how to deal with a new pregnancy, reproductive life plan, and additional health benefits from using contraception.
  3. A tiered effectiveness chart of available contraceptives
  4. A box of contraceptive models
  Interventions: Other: Structured contraceptive counseling

INTERVENTIONS:
Other: Structured contraceptive counseling — 1. Educational video - healthcare providers (Medical doctors and nurse-midwives)present available contraceptives that could be used after delivery, with emphasis on effectiveness, how they should be used, mechanism of action and health benefits.
  2. The four key questions are to be asked to all pregnant women to make them reflect on factors that highly affects choice of contraceptives.
  3. A tiered effectiveness chart will be used to visualize the effectiveness of different contraceptives, and guide the prospective user in her choice depending on the answers to the key questions
  4. The box of contraceptive models are used for the prospective user to inspect, hold, feel the different contraceptives, as this has been shown to decrease fear regarding specific methods.

SUMMARY:
Unintended pregnancy is common among women of fertile age, and also among those who have recently given birth. A Swedish study has shown that about 7.7% experience a new pregnancy, and that 2.5% will have an abortion between 12-24 months from childbirth.

This is a prospective observational intervention study, aiming to evaluate the effects of structured contraceptive counseling during pregnancy on uptake of contraception postpartum and more specifically on long-acting reversible contraceptive methods, and to identify and explore the provider's and patient's experiences of structured contraceptive counseling during pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older, gestational week 30 or more, need for contraception 6 months or more after delivery

Exclusion Criteria:

- Language barrier that affects participation when an interpreter is not available, assisted fertilization, planned sterilization of partner, use of contraception for other purposes than pregnancy prevention.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2022-11-19 (Actual); Primary Completion 2025-06-19 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Difference in proportions of LARC use 6 months postpartum among women receiving structured contraceptive counseling compared to standard care during pregnancy. | 6 months post partum
  Percentage

SECONDARY OUTCOMES:
New pregnancy | 6, 12, 18, and 24 months postpartum
  Categorical (yes/no)
Outcome of new pregnancy | 6, 12, 18, nd 24 months postpartum
  Categorical (yes/no) for planing to keep; kept; misscarriage; ectopic pregnancy; planning abortion; had an abotion

CONTACTS AND LOCATIONS:
Overall Officials: Niklas Envall, PhD, Principal Investigator — Dalarna University
Locations (4):
- Sweden (4):
  - Health Care Region Dalarna, Falun
  - Health Care Region Värmland, Karlstad
  - Health Care Region Örebro Län, Örebro
  - Health Care Region Uppsala, Uppsala

IPD SHARING:
Plan to Share IPD: Yes
Upon request, de-identified data might be shared with other researchers that share the purpose of this trial